CLINICAL TRIAL: NCT03899441
Title: Does Multimedia Perioperative Teaching Improve Patient Experience in the Treatment of Endometrial Cancer
Brief Title: Multimedia Aid Gynecologic Counseling and Consent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1821
Record Dates: First submitted 2019-03-01; First posted 2019-04-02 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Endometrium Cancer; Sentinel Lymph Node; Perioperative/Postoperative Complications
Keywords: multimedia, video teaching
MeSH Terms: conditions — Endometrial Neoplasms; Postoperative Complications | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control arm will have pre-operative teaching from their physician and sign consent for surgery, as is the current standard of care at the investigators' institution.
- Video arm (Experimental): Patients in the intervention arm will watch two short animated video about minimally-invasive endometrial cancer surgery followed by focused pre-operative teaching from their physician. They will then sign consent for surgery.
  Interventions: Other: Video

INTERVENTIONS:
Other: Video — Two short animated videos - one that reviews minimally-invasive surgery and sentinel lymph node mapping and biopsy for endometrial cancer treatment. This video as reviews possible complications. The second video reviews peri-operative instructions.
  Arms: Video arm

SUMMARY:
This is an interventional trial to introduce two short animated videos into preoperative counseling/consent and to compare patient comprehension and satisfaction with a multimedia approach compared to standard of care currently. The investigators anticipate that patients will retain more information about their surgery and peri-operative care and will be more satisfied with a multimedia approach.

DETAILED DESCRIPTION:
The investigators plan a pilot study where patients will be randomized to receiving standard consent and teaching prior to their planned surgery for endometrial cancer or standard consent and multimedia video aid with targeted teaching. This video will be an adjunct to the standard consent process and supplement the pre and post-operative teaching that is currently not formalized. The primary outcome is patient satisfaction. The secondary outcomes include patient understanding and physician satisfaction. The investigators hypothesize that patients will be more satisfied when their consent for surgery is done in conjunction with this multimedia aid.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Has diagnosis of endometrial cancer
* Planned minimally invasive surgical treatment with hysterectomy and sentinel lymph node biopsy

Exclusion Criteria:

* Non-English speaking
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 1 day (assessed at first visit)
  Patient satisfaction with the clinic visit (either new patient visit where they are consented for surgery or a pre-operative visit). Patient satisfaction will be measured using two survey tools: a single question to assess global satisfaction with the clinic visit (on a scale from 1-10) and an 8 question validated satisfaction survey (Client Satisfaction Questionnaire-8 or CSQ-8). Patient satisfaction will be compared between the control and intervention groups. For the single question satisfaction question, answers are on a scale from 1-10, the higher numbers indicating higher satisfaction. The CSQ8 survey contains 8 questions that all have answers ranging from 1 to 4, with higher numbers indicating higher satisfaction.

SECONDARY OUTCOMES:
Patient comprehension | 6-8 weeks (assessed at 3 time points - first clinic visit, inpatient at time of surgery, and at follow-up visit 4-6 weeks after surgery)
  Patient comprehension (of the surgery, its complication, and peri-operative instructions) will be measured using a 9 question survey developed by the study investigators. This survey was developed to assess patient understanding on key information reviewed either in the study videos or by physicians during pre-operative counseling. Patient comprehension will be assessed at three different time points (using the same survey) to compare comprehension immediately after watching the video or undergoing standard physician counseling and again during the patient's hospital stay and at the follow-up visit. Comprehension scores will be compared between the control and intervention groups. The comprehension surveys questions will all be awarded points for correct answers, with higher answers indicating more comprehension of topics relating to the surgery.
Physician satisfaction | 1 day (assessed at first visit)
  Physician satisfaction with new patient or pre-operative visit. Physician satisfaction will be measured using a single question to assess global satisfaction with the clinic visit (on a scale from 1-10, with higher numbers indicating higher satisfaction).
Visit length | 1 day (assessed during first visit)
  Time of new patient or pre-operative visit. The length of visits will be recorded (from the time the physician first enters the patient room until the visit is complete and the patient is leaving the clinic room). Appointment times will be compared between the control and intervention group, for pre-operative visits and new patient visits.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tucker, MD, Principal Investigator — UNC Hospital
Locations (1):
- Univeristy of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No